CLINICAL TRIAL: NCT01631409
Title: Estimation of the Long Term Effectiveness of Routine Use of Cardiac Shock Wave Therapy in the General System of Noninvasive, Invasive, and Surgical Treatment of Ischemic Heart Disease in the Conditions of a Large General City Hospital
Brief Title: Estimation of the Long Term Effectiveness of Routine Use of Cardiac Shock Wave Therapy
Acronym: CSWTSPB40
Status: Withdrawn | Type: Observational
Why Stopped: The study has been withdrawn due to organizational problems
Sponsor: City Hospital No 40, Saint Petersburg, Russia (Other)
Responsible Party: Sponsor
Other Study IDs: CSWT City Hosp No 40, SPB, Ru
Record Dates: First submitted 2012-06-24; First posted 2012-06-29 (Estimated); Last update posted 2014-04-08 (Estimated); Status verified 2014-04

CONDITIONS: Coronary Heart Disease (CHD)
Keywords: clinical research; coronary heart disease; cardiac shock wave therapy; ischemic heart disease; myocardial revascularization; observational research; prospective research
MeSH Terms: conditions — Coronary Disease; Myocardial Ischemia | interventions — Simvastatin; Aspirin; isosorbide-5-mononitrate; Atenolol; Enalapril; Nitroglycerin; Enalaprilat; Amlodipine; Passive Cutaneous Anaphylaxis; Coronary Artery Bypass

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes

GROUPS / COHORTS (7):
- Cohort 0: Cohort 0 is allocated for the following two patient groups:
  1. The patients with suspicion of angina although in whom the thorough investigation has not revealed CHD and the pain syndrome has been received the extracardiac interpretation (e.g. vertebral osteochondrosis, left side humeroscapular periarthritis, herpes zoster, intercostal neuralgia Tietze syndrome etc.)
  2. The patients with subclinical manifestation of coronary atherosclerosis without angina (Class 0 angina, here and further is according to the Canadian Cardiovascular Society Angina Classification). This subgroup of the patients is recommended the proper diet, life style modification, lipid targeting medications in some cases, and no antianginal treatment.
  Interventions: Other: Treatment of CHD risk factors
- Cohort I: Represents patients with Class 1 angina, who receive OMT.
  Interventions: Drug: Aspirin, Isosorbide mononitrate, Atenolol, Enalapril.
- Cohort II: Comprises the patients with Class 2-4 angina, they are on MAAMT. The cohort is further divided in two groups:
  1. The patients for whom MAAMT is effective.
  2. The patients for whom MAAMT is not effective or not sufficiently effective, although those patients have not received any invasive, surgical or CSWT interventions yet.
  They are those patients who then form cohorts III-VI.
  Interventions: Drug: Aspirin, Isosorbide mononitrate, Atenolol, Enalapril.
- Cohort III: Consists of patients already received PCA. They also continue various MAAMT.
  Interventions: Procedure: PCA
- Cohort IV: Includes the patients after CABG. They also are on various MAAMT.
  Interventions: Procedure: CABG
- Cohort V: Incorporates the patients who have already underwent CSWT. They also receive individualized MAAMT.
  Interventions: Device: Cardiospec
- Cohort VI: The cohort is composed of the patients who for various reasons have not been exposed to any intervention except MAAMT and continue to be on it.
  The algorithm of the cohort formation is graphically demonstrated in the Diagram "The logic tree of the cohort formation" (see the link at the bottom of the protocol).
  Interventions: Drug: Aspirin, Isosorbide mononitrate, Atenolol, Enalapril

INTERVENTIONS:
Other: Treatment of CHD risk factors — Smoking cessation, low fat diet, body weight control, physical exercise program, and in some cases lipid-lowering medications, e.g. 3-hydroxy-3-methylglutaric acid-coenzyme A (HMG-CoA) reductase inhibitors, e.g. Simvastatin.
  Other Names: Life style modification, sports, Zocor.
  Groups: Cohort 0
Drug: Aspirin, Isosorbide mononitrate, Atenolol, Enalapril. — In the course of optimal medical treatment of Cohort I patient the life style modification is combined with one group of antianginal medications (e.g. Nitrates, Beta-blockers, ACE inhibitors, Calcium antagonists) and lipid-lowering drugs (e.g. HMG-CoA reductase inhibitors).
  Other Names: Halfprin 81, Nitrostat, Monoket, Tenormin, Vasotec, Norvasc.
  Groups: Cohort I
Drug: Aspirin, Isosorbide mononitrate, Atenolol, Enalapril. — In the course of maximal antianginal medical therapy a Cohort II patient is provided with more than one group of antianginal medications (e.g. Nitrates, Beta-blockers, ACE inhibitors, Calcium antagonists) combined with lowering-lipid drugs (e.g. HMG-CoA reductase inhibitors).
  Other Names: Nitrostat, Monoket, Tenormin, Vasotec, Norvasc.
  Groups: Cohort II
Procedure: PCA — Percutaneous coronary angioplasty
  Other Names: e.g. coronary stenting
  Groups: Cohort III
Procedure: CABG — Coronary artery bypass grafting
  Other Names: coronary artery bypass surgery
  Groups: Cohort IV
Device: Cardiospec — Cardiac shock wave therapy is implemented by device Cardiospec manufactured by Medispec Ltd.
  Other Names: noninvasive cardiac revascularization
  Groups: Cohort V
Drug: Aspirin, Isosorbide mononitrate, Atenolol, Enalapril — In the course of maximal antianginal medical therapy a Cohort VI patient is provided with more than two groups of antianginal medications (e.g. Nitrates, Beta-blockers, ACE inhibitors, Calcium antagonists) combined with lowering-lipid drugs (e.g. HMG-CoA reductase inhibitors).
  Other Names: Halfprin 81, Nitrostat, Monoket, Tenormin, Vasotec, Norvasc.
  Groups: Cohort VI

SUMMARY:
This study is dedicated to determination of the long term effectiveness of coronary heart disease (CHD) treatments - cardiac shock wave therapy (CSWT) in comparison with other kinds of medical and surgical treatment. For that purpose the investigators will observe the patients with CHD who enrolled in this study in their routine course of treatment. But the investigators will not interfere with the patient treatment. Each participant will be followed-up for five years. The collected data will allow to determine if the particular method, CSWT, could really make any additional contribution to the more traditional methods of CHD treatment and if the CSWT is only temporarily effective or could exert the long term effect as well.

DETAILED DESCRIPTION:
This study has been designed and is conducted in accordance with the requirements of Helsinki Declaration, 6th edition, STROBE Statement, CONSORT 2010 Statement, and the State Standard of the Russian Federation "Guidelines for Clinical Investigations of Medical Devices" (ГОСТ Р ИСО 14155 - 2008), which is authentic to International Standards Organization standard 141555 - 2003.

According to the American Heart Association (AHA) 2011 report Russia leaves behind all other countries in the coronary heart disease mortality rate. This particularly means that the current methods of CHD treatment, namely: (1) optimal medical treatment (OMT), which includes intensive lifestyle and pharmacological management, (2) maximal antianginal medical therapy (MAAMT), which includes the employment of at least two classes of anti-ischemic therapies, (3) percutaneous coronary angioplasty (PCA), and (4) coronary artery bypass grafting (CABG) are not satisfactory enough in the concrete conditions of Russia. This indicate the urgent necessity of search for the alternative methods of CHD treatment. One of those methods is cardiac shock wave therapy.

The method of CSWT is not that new. The first publication is dated back to 1999. Since then a score of various in vivo as well clinical investigations has been conducted up to phase III. As a result, it has been demonstrated that (1)the method is practically safe and well-tolerated, and (2)it effectively alleviates angina and improves ECG, ECHO, and cardiac nuclear tests. Meanwhile, it is still not clear: (1) how long the remission lasts, (2)if CSWT exerts any influence on such basic health indicators as life span and reduction of major cardiovascular (CV) events like myocardial infarction (MI), (3)the place of CSWT in the overall system of conservative and surgical treatment of CHD, and (4)the long term effect of combined employment of CSWT with invasive and surgical modalities.

One of the causes of the such a state of things is the form in which CSWT research so far has been conducted, namely, the clinical trial. The high cost of that type of investigations precludes long-term follow-up. Besides, the desire to make the experimental and control group more homogeneous in the parallel design using multiple inclusion/exclusion criteria dramatically decreases sample representativeness. The observational design is mostly free of the above-mentioned shortcomings and in some instances allows to obtain important results which even theoretically are not accessible for investigations with strict control and randomization because of ethical and pragmatic considerations.

The aim of this study is to estimate the long term effectiveness of routine use of cardiac shock wave therapy in the general system of noninvasive, invasive, and surgical treatment of ischemic heart diseases in the conditions of a large general city hospital. The study will be conducted in the City Hospital No 40, Saint Petersburg, Russia (about the hospital see the link at the bottom of the protocol). It is a more than thousand bed general hospital. There are 55 thousand adults live within its zone of responsibility. From those there are approximately two thousand patients with CHD.

The algorithm of treatment selection in the hospital. The treatment of all patients begins from OMT. When OMT is not effective MAAMT is administered. The medical therapy is conducted strictly individually. When MAAMT fails the patient is offered PCA or CABG. That is, the general ideology of CHD therapy in the hospital follows the conventional international guidelines. CSWT is offered mostly in two cases: (1)when the patient refuses to undergo PCA or CABG, (2)when PCA or CABG are contraindicated for the patient. That is CSWT is factually used as the second line, reserve method.

In the hospital, CSWT is routinely employed for three years in correspondence with the prevailed international scheme: 3 sessions a week every first week for three consecutive months, 9 sessions altogether according to the guidelines approved by the First deputy of Saint Petersburg health care committee chairman. The CSWT is implemented by device Cardiospec manufactured by Medispec Ltd., headquarters in Germantown, MD, USA. The zone of reversed myocardial ischemia for CSWT application is determined by ECHO.

For the current study there will be formed seven observational cohorts (0-VI) by both diagnoses and interventions. The algorithm of the cohort formation in the current study is graphically demonstrated in the Diagram (see the link at the bottom of the protocol). The enrollment in the study will continue for 3 year. Taking into consideration the current CHD morbidity rate in the region 6,5‰, that allows to expect an additional one thousand patients for the investigation. Each participant will follow-up for five years. So the total length of the study is eight years.

ELIGIBILITY:
Inclusion Criteria:

1. Age 18 years and older.
2. Diagnosed or suspected CHD.
3. Willingness to participate in the study.

Exclusion Criteria:

* Inability of a patient to make an independent decision on participation in the study because of intellectual decline (article 29 of Helsinki Declaration)

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: There are 55 thousand adults live within the zone of responsibility of the hospital. From those there are approximately 2 thousand patients with CHD.
Sampling Method: Non-Probability Sample
Enrollment: 0 (Actual)
Dates: Start 2013-09; Primary Completion 2021-09 (Estimated); Study Completion 2021-09 (Estimated)

PRIMARY OUTCOMES:
Outcome: death | within three years after the enrolment
  the detailed circumstances and diagnose are determined by documents
Outcome: major cardiovascular complications | within three years after the enrolment
  the detailed circumstances and diagnose are determined by documents

SECONDARY OUTCOMES:
The number of hospitalizations | within three years after the enrolment
  determined by documents
The number of hospitalization days | within three years after the enrolment
  determined by documents

CONTACTS AND LOCATIONS:
Overall Officials: Sergey G Scherbak, MD, Prof., Study Director — City Hospital No 40, Saint Petersburg, Russia; Dmitriy G Lisovetz, MD, CMedSc, Principal Investigator — City Hospital No 40, Saint Petersburg, Russia

REFERENCES:
- See also: About the City Hospital No40, Saint Petersburg, Russia see its Wikipedia page — http://en.wikipedia.org/wiki/City_hospital_No_40,_Saint_Petersburg,_Russia